CLINICAL TRIAL: NCT04197427
Title: Determination of the Safety and Efficacy of a Novel Oral Rinse on Oral Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: You First Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SW-101-19
Record Dates: First submitted 2019-12-04; First posted 2019-12-13 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Plaque; Gingivitis
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Experimental Oral Rinse (Experimental): In this arm the test article,oral rinse, a proprietary formulation of agents including xylitol, Caffeine, Essential oils, Monk fruit extract, which can reduce the plaque formation Subjects rinse twice a day with 10 mL of the oral rinse for 2 minutes for 30 days.
  They will note, in the daily oral hygiene diary, the date and time of brushing and rinsing.
  Interventions: Device: Experimental Oral Rinse
- Placebo Oral Rinse (Placebo Comparator): This arm will use a placebo with out the active ingredients same way the experimental arm do.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Experimental Oral Rinse — Experimental Oral Rinse is a proprietary formulation of GRAS ingredients
  Arms: Experimental Oral Rinse
Device: Placebo — Placebo formulation without the active ingredients
  Arms: Placebo Oral Rinse

SUMMARY:
Since over 50% of the US population have gingivitis, mouthrinses serve as a valuable adjunct to brushing and flossing. The primary objective is to determine the effectiveness of the oral rinse in reducing plaque and gingivitis and improve a patient's breath

DETAILED DESCRIPTION:
This clinical study design is a randomized, double-blind, single-treatment, parallel design with a placebo as the control. Following a screening exam, the duration of the trial will be 1 month. Oral examinations will occur at Visit 1 (baseline), and Visit 2 (4 weeks post screening). Also, at these visits, subjects will be asked keep a diary for the one month and their thoughts about the effect of the mouthrinse on their breath and their mouth feeling of "freshness". They will also be asked about the taste and consistency of the mouth rinse. Plaque accumulation will be measured by the Turesky modification of the Quigley-Hein method of quantifying plaque formulation (PI). Gingival health will be measured using the Modified Gingival Index (MGI)

ELIGIBILITY:
Inclusion Criteria:

* Subject has read, signed and received a copy of the Informed Consent and HIPAA authorization prior to study initiation.
* Subject is able to follow verbal and/or written instructions, perform oral hygiene procedures and return to the test facility for specified study examinations.
* Subject is between the ages of 18 and 75 years inclusive.
* Subject will not have professional cleaning during the study.
* Subject has no history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test drug, as determined by the Principal Investigator.
* Subject has a minimum of 12 natural teeth.
* Subject agrees to refrain from the use of any oral rinse, toothpaste or dentifrice other than the Aim® Fluoride toothpaste and study rinse provided on Visit 1 for the duration of the study.
* Subject agrees to refrain from the use of other oral care products not supplied by the study center
* Subject agrees to be compliant with study procedures.
* Females of childbearing potential agree to use an adequate method of birth control and agree to pregnancy

Exclusion Criteria:

* Subject has read, signed and received a copy of the Informed Consent and HIPAA authorization prior to study initiation.
* Subject is able to follow verbal and/or written instructions, perform oral hygiene procedures and return to the test facility for specified study examinations.
* Subject is between the ages of 18 and 75 years inclusive.
* Subject will not have professional cleaning during the study.
* Subject has no history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test drug, as determined by the Principal Investigator.
* Subject has a minimum of 12 natural teeth.
* Subject agrees to refrain from the use of any oral rinse, toothpaste or dentifrice other than the Aim® Fluoride toothpaste and study rinse provided on Visit 1 for the duration of the study.
* Subject agrees to refrain from the use of other oral care products not supplied by the study center
* Subject agrees to be compliant with study procedures.
* Females of childbearing potential agree to use an adequate method of birth control and agree to pregnancy testing at the first and second visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the oral rinse in reducing plaque | 4 weeks
  Plaque accumulation will be measured by the Turesky modification of the Quigley-Hein method of quantifying plaque formulation (PI).
Effectiveness of the oral rinse in reducing gingivitis | 4 weeks
  Gingival health will be measured using the Modified Gingival Index (MGI)
Effectiveness of the oral rinse in improving a patient's breath | 4 weeks
  Subjects will be asked keep a diary for one month and their thoughts about the effect of the mouthrinse on their breath and their mouth feeling of "freshness",

SECONDARY OUTCOMES:
Safety evaluation of the test Oral Rinse | 4 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontics and Endodontics,School of Dental Medicine, University at Buffalo, SUNY, Buffalo, New York, United States